CLINICAL TRIAL: NCT06768320
Title: Parent Toddler Obesity Study (PTOS)
Brief Title: Treating Toddler Obesity by Treating the Parent/Caregiver Obesity With Weight Loss Medications
Acronym: PTOS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficult to recruit. an unexpected result is the easy availability of GLP 1 medication to the general public.
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB 5240207
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Weight Loss; Obesity, Childhood; Obesity
MeSH Terms: conditions — Weight Loss; Pediatric Obesity; Obesity | interventions — Phentermine; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Lomaira (Active Comparator): Participants will receive Lomaira 8mg for 12 weeks and off 12 weeks, will restart at week 24 for 12 weeks one tablet per day 30 minutes before a meal.
  Interventions: Drug: Lomaira 8Mg Tablet
- Placebo (No Intervention): Participants will receive Placebo for 12 weeks and off 12 weeks, will restart at week 24 for 12 weeks one tablet per day 30 minutes before a meal.

INTERVENTIONS:
Drug: Lomaira 8Mg Tablet — 8 mg tablet up to three times a day
  Arms: Active Lomaira

SUMMARY:
The purpose of this study is to treat toddler obesity by improving the toddler nutritional environment. Parents will participate in a free internet nutrition program and may also take obesity medication. These measures may improve the parental nutritional environment and in turn, improve the toddler nutritional environment as well.

DETAILED DESCRIPTION:
Fifty parent or caregiver and toddler teams will be enrolled in a 37 week study in which the parents or caregivers will be randomized to receive either an obesity drug or a placebo, while simultaneously enrolled in the Full Plate Living lifestyle program. Study eligibility and ongoing participation will be assessed by lab results, biometric measurements and nutrition questionnaires to monitor the impact of diet and medication on the parental dietary environment. Toddler body mass index (BMI) will be calculated at study inception and completion to assess potential impact on the toddler dietary environment. Teaching will be provided to parents on healthy dietary choices, adequate sleep and stress control.

ELIGIBILITY:
Inclusion Criteria: Adults

* Self-identify as being of Hispanic/Latino or African American ethnicity
* BMI ≥30 with a stable weight (no more than 5% variation during the previous 3 months) and an agreement not to initiate any other weight loss
* HbAlc ≤ 6.4
* Fluent in written and spoken English

Exclusion Criteria: Adult

* Current cancer treatment
* Have been treated with prescription drugs that promote weight loss (for example, liraglutide [Saxenda™], orlistat [Xenical®], phentermine Adipex®], phentermine/topiramate [Qsymia™], semaglutide 2.4 mg [Wegovy™], tirzepatide [Zepbound™], bupropion/naltrexone [Contrave™], phentermine [Lomaira™] or similar other weight loss medications including over-the-counter (OTC) medications (for example, Alli®). Use of obesogenic medications (including but not limited to steroids, haloperidol, clozapine, risperidone, olanzapine, amitriptyline, imipramine, paroxetine, and lithium) which cannot be substituted or stopped
* History of drug or alcohol abuse
* Nursing or planning to become pregnant in the next 10 months
* Unwilling to use accepted standards of birth control if female and before menopause age. (i.e. IUD, birth control pills/injections, tubal or vas deferens ligation) during the study and for 30 days after the study is completed. Condoms or rhythm methods are not sufficient.

Inclusion Criteria: (Toddler)

* Self-identify as being of Hispanic/Latino or African American ethnicity
* BMI ≥ 95th percentile for age, gender and height
* Age 12 to 36 months of age
* Spends at least half of its awake time per day with the P/OCG who is the consenting adult and who provides at least half of the toddler's diet on that day

Exclusion Criteria (Toddler)

* Current cancer treatment
* Use of obesogenic medications (including but not limited to steroids, haloperidol, clozapine, risperidone, olanzapine, amitriptyline, imipramine, paroxetine, and lithium) which cannot be substituted or stopped
* Genetic disorders and/or physical or mental handicaps that would limit participation in the study and/or the lifestyle intervention
* Any special dietary or exercise requirements
* Any established chromosome abnormalities that might be associated with obesity

Ages: 12 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change in Toddler's Body Mass index (BMI) percentile at week 37 | Change between baseline visit and final study visit at week 37
  Toddler BMI will be measured at enrollment and at final study visit week 37. BMI will be calculated using the InBody Scale. This is a composite measurement consisting of height and weight.
Change in parent's Body Mass index (BMI) at week 37 | Change between baseline visit and final study visit at week 37
  Adults BMI will be measured at enrollment and at final study visit week 37. BMI will be calculated using the InBody Scale. This is a composite measurement consisting of height and weight.

CONTACTS AND LOCATIONS:
Overall Officials: Warren C Peters, MD, Principal Investigator — Loma Linda University (School of Public Health)
Locations (2):
- United States (2):
  - Loma Linda University, Loma Linda, California
  - Nutrition Research Center, Loma Linda, California

IPD SHARING:
Plan to Share IPD: No
No formal plans